CLINICAL TRIAL: NCT05884814
Title: Timing of Resistance Exercise, Glucose Control and Exercise Adaptations in People With Type 1 Diabetes: a Randomised-controlled Trial
Brief Title: Timing of Resistance Exercise in Type 1 Diabetes
Acronym: T-REX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dasman Diabetes Institute (Other)
Responsible Party: Principal Investigator, Dr. Ebaa Al Ozairi, Chief Medical Officer, Dasman Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RA HM-2023-009
Record Dates: First submitted 2023-05-10; First posted 2023-06-01 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Type 1 Diabetes
Keywords: exercise; circadian rhythm; glucose control; muscle; strength
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Intervention Model Description: 1:1:1 parallel group design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Habitual physical activity
  Interventions: Behavioral: Habitual physical activity levels
- Morning exercise (Active Comparator): Exercise training between 6-10am
  Interventions: Behavioral: Morning exercise
- Afternoon exercise (Active Comparator): Exercise training between 4-8pm
  Interventions: Behavioral: Afternoon exercise

INTERVENTIONS:
Behavioral: Morning exercise — Between 6-10am participants will attend the gym and perform 10 min of warm up exercise, 3 sets of 7 resistance exercises ( leg press, calf press, leg curl, chest press, lateral raise, seated row and plank)
  Arms: Morning exercise
Behavioral: Afternoon exercise — Between 4-8pm participants will attend the gym and perform 10 min of warm up exercise, 3 sets of 7 resistance exercises ( leg press, calf press, leg curl, chest press, lateral raise, seated row and plank)
  Arms: Afternoon exercise
Behavioral: Habitual physical activity levels — Participants will be asked to maintain their normal activity levels
  Arms: Control

SUMMARY:
The aims of the current study are

1. to compare the effects of acute morning and afternoon resistance exercise on blood glucose levels in people with type 1 diabetes.
2. to compare the effects of morning and afternoon resistance exercise training on cardiometabolic health outcomes in people with type 1 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Physician confirmed type 1 diabetes for at least 1 year
* Stable insulin therapy for 3 months prior to the study

Exclusion Criteria:

* BMI of 45 or higher
* BP of 160/100mmHg or higher
* autonomic neuropathy
* severe proliferative retinopathy
* joint or limb injuries preventing weight-bearing activity
* autonomic neuropathy
* severe proliferative retinopathy
* any other medical condition that prevents participants from exercising safely.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in muscle strength | Change from baseline to 12 weeks
  Sum of one repetition maximum for the 7 resistance exercise
Change in interstitial glucose time in range | Change from 6 hours before (baseline) to 6 hours after (post-exercise) an exercise training session
  Interstitial glucose time in range (3.9-10mmol/L) measured via continuous glucose monitoring

SECONDARY OUTCOMES:
Change in appendicular skeletal muscle mass | Change from baseline to 12 weeks
  Measured by DEXA
Change in whole body fat mass | Change from baseline to 12 weeks
  Measured by DEXA
Change in physical function | Change from baseline to 12 weeks
  Measured by the short performance physical battery
Change in HbA1c | Change from baseline to 12 weeks
  HbA1c concentration
Change in interstitial glucose average | Change from 6 hours before (baseline) to 6 hours after (post-exercise) an exercise training session
  Interstitial average glucose measured via continuous glucose monitoring
Change in interstitial glucose variability | Change from 6 hours before (baseline) to 6 hours after (post-exercise) an exercise training session
  Interstitial glucose variability measured via continuous glucose monitoring
Change in interstitial glucose time in hypoglycaemia | Change from 6 hours before (baseline) to 6 hours after (post-exercise) an exercise training session
  Interstitial glucose time in range (<3.9mmol/L) measured via continuous glucose monitoring
Change in interstitial glucose time in hyperglycaemia | Change from 6 hours before (baseline) to 6 hours after (post-exercise) an exercise training session
  Interstitial glucose time in range (>10mmol/L) measured via continuous glucose monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No